CLINICAL TRIAL: NCT01614470
Title: A Phase 3, Two-Part, Randomized, Double-Blind, Placebo-Controlled, Crossover Study With an Open-Label Period to Evaluate the Efficacy and Safety of Ivacaftor in Subjects With Cystic Fibrosis Who Have a Non-G551D CFTR Gating Mutation
Brief Title: Study of Ivacaftor in Subjects With Cystic Fibrosis (CF) Who Have a Non-G551D CF Transmembrane Conductance Regulator (CFTR) Gating Mutation
Acronym: KONNECTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX12-770-111
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1: Ivacaftor First, Then Placebo (Experimental): Ivacaftor 150 milligram (mg) tablet orally twice daily for 8 weeks in treatment period 1 followed by placebo matched to ivacaftor tablet orally twice daily for 8 weeks in treatment period 2. Washout out period of 4 to 8 weeks was maintained between each treatment period.
  Interventions: Drug: Ivacaftor; Drug: Placebo
- Part 1: Placebo First, Then Ivacaftor (Experimental): Placebo matched to ivacaftor tablet orally twice daily for 8 weeks in treatment period 1 followed by ivacaftor 150 mg tablet orally twice daily for 8 weeks in treatment period 2. Washout out period of 4 to 8 weeks was maintained between each treatment period.
  Interventions: Drug: Ivacaftor; Drug: Placebo
- Part 2: Ivacaftor (Experimental): Ivacaftor 150 mg tablet orally twice daily for 16 weeks.
  Interventions: Drug: Ivacaftor

INTERVENTIONS:
Drug: Ivacaftor — 150 mg tablet, oral use, administered twice a day (q12h)
  Other Names: Kalydeco; VX-770
Drug: Placebo — oral use, administered twice a day (q12h)
  Arms: Part 1: Ivacaftor First, Then Placebo; Part 1: Placebo First, Then Ivacaftor

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ivacaftor in subjects with cystic fibrosis (CF) who have a non-G551D cystic fibrosis transmembrane regulator (CFTR) gating mutation (any one of the following CFTR mutations: G178R, G551S, S549N, S549R, G970R, G1244E, S1251N, S1255P, or G1349D).

DETAILED DESCRIPTION:
Ivacaftor is the first CFTR modulator to show an improvement in CFTR function and clinical benefit in subjects with CF. Results from Phase 3 studies (VX08-770-102 [Study 102] [NCT00909532] and VX08-770-103 [Study 103] [NCT00909727]) showed that ivacaftor is effective in the treatment of subjects with CF who have the G551D-CFTR mutation, as evidenced by sustained improvements in CFTR channel function (measured by reduction in sweat chloride concentration) and corresponding substantial, durable improvements in lung function, pulmonary exacerbations, respiratory symptoms, and weight gain. Ivacaftor was also well tolerated, as evidenced by the rates and reasons for premature discontinuation and results of safety assessments.

Ivacaftor (Trade Name Kalydeco; 150 mg tablets) was initially approved in the United States for the treatment of CF in subjects 6 years of age and older who have a G551D mutation in the CFTR gene.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF
* At least 1 allele of the following CFTR gating mutations: G178R, S549N, S549R, G551S, G970R, G1244E, S1251N, S1255P, G1349D
* Percent predicted forced expiratory volume in 1 second (FEV1) greater than or equal to (>=) 40 percent (%) predicted normal for age, sex, and height
* 6 years of age or older
* Minimum weight of 15 kilogram (kg) at screening
* Females of childbearing potential must not be pregnant
* Willing to comply with contraception requirements

Exclusion Criteria:

* G551D-CFTR mutation on at least 1 allele
* History of any illness or condition that might confound the results of the study or pose an additional risk in administering ivacaftor to the subject
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before the first dose of study drug
* History of solid organ or hematological transplantation
* History of alcohol, medication or illicit drug abuse within 1 year before the first dose of study drug
* Ongoing participation in another therapeutic clinical study or prior participation in an investigational drug study within 30 days before screening
* Use of inhaled hypertonic saline treatment
* Use of any inhibitors or inducers of cytochrome (CYP) P450 3A
* Evidence of cataract or lens opacity at screening

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine De Boeck, MD, PhD, Principal Investigator — University of Leuven
Locations (12):
- United States (8):
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Houston, Texas
- Leuven, Belgium
- France (3):
  - Lyon
  - Montpellier
  - Paris

RESULTS

PARTICIPANT FLOW:
Period: Part 1: Treatment Period 1 (8 Weeks)
Arm/Group | Part 1: Ivacaftor First, Then Placebo | Part 1: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 20 | 19 | 0
Completed | 18 | 18 | 0
Not Completed | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Need to extend washout period | 1 | 1 | 0
Period: Part 1: Washout Period (4 to 8 Weeks)
Arm/Group | Part 1: Ivacaftor First, Then Placebo | Part 1: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 18 | 18 | 0
Completed | 18 | 18 | 0
Not Completed | 0 | 0 | 0
Period: Part 1: Treatment Period 2 (8 Weeks)
Arm/Group | Part 1: Ivacaftor First, Then Placebo | Part 1: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 18 | 18 | 0
Completed | 18 | 18 | 0
Not Completed | 0 | 0 | 0
Period: Part 2: Open-label Period (16 Weeks)
Arm/Group | Part 1: Ivacaftor First, Then Placebo | Part 1: Placebo First, Then Ivacaftor | Part 2: Ivacaftor
Started | 0 | 0 | 36
Completed | 0 | 0 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) was defined as all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Ivacaftor First, Then Placebo | Part 1: Placebo First, Then Ivacaftor | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (13.25) | 21.7 (12.92) | 22.8 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through Week 8
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male subjects 18 years and older and female subjects 16 years and older. The Wang standard was used for male subjects aged 6 to 17 years and for female subjects aged 6 to 15 years. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during study Part 1.
Time Frame: Part 1: Baseline (pre-dose Day 1), Week 8
Population: FAS for Part 1: all randomized subjects who received at least 1 dose of study drug (ivacaftor or placebo). Here, "n" signifies those subjects who were evaluable for this measure at given time point for each group, respectively.
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Groups:
- Part 1: Ivacaftor: Ivacaftor 150 mg tablet orally twice daily for 8 weeks in either treatment period 1 or treatment period 2.
- Part 1: Placebo: Placebo matched to ivacaftor tablet orally twice daily for 8 weeks in either treatment period 1 or treatment period 2.
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo
Number analyzed (Participants) | 38 | 37
percent predicted of FEV1
  Baseline (n=38, 37) | 76.3659 (20.33450) | 79.3361 (20.83991)
  Change Through Week 8 (n=37, 37) | 8.1308 (9.94676) | -5.8738 (7.23722)
Statistical Analysis 1: Comparison: Part 1: Ivacaftor vs Part 1: Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Least squares (LS) mean difference = 10.6780, 95% CI 2-sided [7.2559 to 14.1000]

2. Secondary Outcome: Part 1: Change From Baseline in Body Mass Index (BMI) at Week 8
Description: BMI was defined as weight in kilogram (kg) divided by height in meters^2 (m^2). Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during study Part 1.
Time Frame: Part 1: Baseline (pre-dose Day 1), Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo
Number analyzed (Participants) | 38 | 37
kg/m^2
  Baseline (n=38, 37) | 22.241 (5.1880) | 22.527 (4.9956)
  Change at Week 8 (n=37, 37) | 0.748 (0.5793) | 0.043 (0.6980)
Statistical Analysis 1: Comparison: Part 1: Ivacaftor vs Part 1: Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS mean difference = 0.6624, 95% CI 2-sided [0.3366 to 0.9881]

3. Secondary Outcome: Part 2: Change From Baseline in Body Mass Index (BMI) at 24 Weeks of Treatment (Week 36 Visit)
Description: BMI was defined as weight in kg divided by height in m^2. Change in BMI over 24 weeks of ivacaftor treatment (from Week 12 [Part 1: Treatment Period 2] through Week 36 [Part 2]) was reported for subjects who received ivacaftor in Part 1: Treatment Period 2 as per planned analysis. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during Part 1: Treatment Period 2.
Time Frame: Baseline (pre-dose Week 12), Week 36
Population: FAS for Part 2: all randomized subjects who received at least 1 dose of study drug (ivacaftor). Only subjects who were randomized to receive ivacaftor during Part 1: Treatment Period 2 were to be analyzed for this measure.
Measure: Mean (Standard Deviation); unit: kg/m^2
Groups:
- Part 1 Treatment Period 2: Ivacaftor, Part 2: Ivacaftor: Ivacaftor 150 mg tablet orally twice daily for 24 weeks (8 weeks in Part 1: Treatment Period 2 and 16 weeks in Part 2).
Arm/Group | Part 1 Treatment Period 2: Ivacaftor, Part 2: Ivacaftor
Number analyzed (Participants) | 18
kg/m^2
  Baseline | 22.222 (6.2919)
  Change at Week 36 | 1.263 (0.7588)

4. Secondary Outcome: Part 1: Change From Baseline in Sweat Chloride Through Week 8
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during study Part 1.
Time Frame: Part 1: Baseline (pre-dose Day 1), Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo
Number analyzed (Participants) | 38 | 37
millimole per liter (mmol/L)
  Baseline (n=38, 37) | 93.37 (18.099) | 94.23 (20.581)
  Change Through Week 8 (n=36, 36) | -55.82 (24.890) | -5.63 (9.833)
Statistical Analysis 1: Comparison: Part 1: Ivacaftor vs Part 1: Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS mean difference = -49.1667, 95% CI 2-sided [-56.9527 to -41.3807]

5. Primary Outcome: Part 2: Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Through 24 Weeks of Treatment (Week 36 Visit)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Hankinson and Wang standards were used to calculate percent predicted FEV1 (for age, gender, and height). The Hankinson standard was used for male subjects 18 years and older and female subjects 16 years and older. The Wang standard was used for male subjects aged 6 to 17 years and for female subjects aged 6 to 15 years. Absolute change in percent predicted FEV1 over 24 weeks of ivacaftor treatment (from Week 12 [Part 1: Treatment Period 2] through Week 36 [Part 2]) was reported for subjects who received ivacaftor in Part 1: Treatment Period 2, as per planned analysis. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during Part 1: Treatment Period 2.
Time Frame: Baseline (pre-dose Week 12), Week 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent predicted of FEV1
Arm/Group | Part 1 Treatment Period 2: Ivacaftor, Part 2: Ivacaftor
Number analyzed (Participants) | 18
percent predicted of FEV1
  Baseline | 74.8375 (19.36754)
  Change Through Week 36 | 13.5307 (10.18174)

6. Secondary Outcome: Part 2: Change From Baseline in Sweat Chloride Through 24 Weeks of Treatment (Week 36 Visit)
Description: Sweat samples were collected using an approved Macroduct (Wescor, Logan, Utah) collection device. A volume of greater than or equal to (>=) 15 microliter was required for determination of sweat chloride. Change in sweat chloride over 24 weeks of ivacaftor treatment (from Week 12 [Part 1: Treatment Period 2] through Week 36 [Part 2]) was reported for subjects who received ivacaftor in Part 1: Treatment Period 2 as per planned analysis. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during Part 1: Treatment Period 2.
Time Frame: Baseline (pre-dose Week 12), Week 36
Population: FAS for Part 2: all randomized subjects who received at least 1 dose of study drug (ivacaftor). Only subjects who were randomized to receive ivacaftor during Part 1: Treatment Period 2 were to be analyzed for this measure. Here "n" signifies those subjects who were evaluable for this measure at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part 1 Treatment Period 2: Ivacaftor, Part 2: Ivacaftor
Number analyzed (Participants) | 18
mmol/L
  Baseline (n=18) | 92.03 (11.468)
  Change Through Week 36 (n=17) | -59.24 (32.566)

7. Secondary Outcome: Part 1: Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through Week 8
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during study Part 1.
Time Frame: Part 1: Baseline (pre-dose Day 1), Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo
Number analyzed (Participants) | 38 | 37
units on a scale
  Baseline (n=38, 37) | 70.61 (17.409) | 74.55 (20.616)
  Change Through Week 8 (n=37, 37) | 12.31 (16.891) | -2.33 (20.648)
Statistical Analysis 1: Comparison: Part 1: Ivacaftor vs Part 1: Placebo; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; LS mean difference = 9.6105, 95% CI 2-sided [4.4874 to 14.7336]

8. Secondary Outcome: Part 2: Change From Baseline in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score Through 24 Weeks of Treatment (Week 36 Visit)
Description: The CFQ-R is a validated patient-reported outcome measuring health-related quality of life for subjects with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. Change in CFQ-R respiratory domain score over 24 weeks of ivacaftor treatment (from Week 12 [Part 1: Treatment Period 2] through Week 36 [Part 2]) was reported for subjects who received ivacaftor in Part 1: Treatment Period 2 as per planned analysis. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug during Part 1: Treatment Period 2.
Time Frame: Baseline (pre-dose Week 12), Week 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part 1 Treatment Period 2: Ivacaftor, Part 2: Ivacaftor
Number analyzed (Participants) | 18
units on a scale
  Baseline | 71.30 (19.526)
  Change Through Week 36 | 11.42 (13.604)

9. Secondary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording/clinical laboratory assessment which occurs during course of study, whether it is considered related to study drug or not. SAE: medical event or condition, which falls into any of following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolonged hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: Part 1: From signing of informed consent up to Week 20
Population: Safety Set for Part 1 included all subjects who received at least 1 dose of study drug (ivacaftor or placebo).
Measure: Number; unit: participants
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo
Number analyzed (Participants) | 38 | 37
participants
  AEs | 28 | 31
  SAEs | 4 | 7

10. Secondary Outcome: Part 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 9
Time Frame: Part 2: Week 20 up to Week 40
Population: Safety Set for Part 2 included all subjects who received at least 1 dose of study drug (ivacaftor).
Measure: Number; unit: participants
Arm/Group | Part 2: Ivacaftor
Number analyzed (Participants) | 36
participants
  AEs | 30
  SAEs | 3

ADVERSE EVENTS:
Time Frame: Part 1: From signing of informed consent up to Week 20; Part 2: Week 20 up to Week 40
Arm/Group | Part 1: Ivacaftor | Part 1: Placebo | Part 2: Ivacaftor
Serious Adverse Events (participants affected / at risk) | 4/38 | 7/37 | 3/36
Other Adverse Events (participants affected / at risk) | 27/38 | 30/37 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ivacaftor (N=38) | Part 1: Placebo (N=37) | Part 2: Ivacaftor (N=36)
Distal Ileal Obstruction Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Appendiceal Mucocoele (Gastrointestinal disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Paranasal Cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 6 | 2
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ivacaftor (N=38) | Part 1: Placebo (N=37) | Part 2: Ivacaftor (N=36)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 7 | 6 | 4
Rhinitis (Infections and infestations) | 3 | 2 | 0
Influenza (Infections and infestations) | 2 | 2 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Lung hyperinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 1 | 2
Fatigue (General disorders) | 2 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Exercise tolerance decreased (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Medical device site reaction (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1
Infusion site thrombosis (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 4
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1
Benign intracranial hypertension (Nervous system disorders) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Pulmonary function test decreased (Investigations) | 0 | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thyroid disorder (Endocrine disorders) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.